CLINICAL TRIAL: NCT02440529
Title: Surgeon-Patient Communication: A Randomized Controlled Trial Evaluating the Impact of an Orthopaedic Related Smoking Cessation Discussion After Fracture Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research staff decision
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Nkemakolam Egekeze, Orthopaedic Researcher, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-248
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Orthopaedic Decision Making
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- (Intervention Group) (Active Comparator): The discussion about how smoking cigarettes impacts patient orthopaedic management plus aid
  Interventions: Behavioral: Intervention
- (Control Group) (Active Comparator): The discussion about how smoking cigarettes impacts patient orthopaedic management.
  Interventions: Behavioral: Verbal Group

INTERVENTIONS:
Behavioral: Intervention — Discussion
  Arms: (Intervention Group)
Behavioral: Verbal Group — Detailed Discussion
  Arms: (Control Group)

SUMMARY:
In this study, the investigators are interested in evaluating the impact of an orthopaedic related smoking cessation discussion after fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 year old or older,
* daily smoker
* inpatient post fracture operation,
* patient that have never received an orthopaedic related smoking cessation discussion

Exclusion Criteria:

* Younger than 18,
* patients unable to provide consent
* patients that suffer from auditory/visual/mental disability requiring another individual as a decision-maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Patient Comprehension | 20 minutes
  Knowledge-Based Question

CONTACTS AND LOCATIONS:
Overall Officials: Nkem Egekeze, MD, Principal Investigator — UMKC DEPT OF ORTHOPAEDIC SURGERY; Jonathan Dubin, MD, Study Director — UMKC DEPT OF ORTHOPAEDIC SURGERY; Karen Williams, PhD, Study Director — UMKC DEPT OF BIOINFORMATICS; Akin Cil, MD, Study Director — UMKC DEPT OF ORTHOPAEDIC SURGERY; Mark Bernhardt, MD, Study Chair — UMKC DEPT OF ORTHOPAEDIC SURGERY; Dane Church, MD, Study Director — UMKC DEPT OF ORTHOPAEDIC SURGERY
Locations (1):
- Truman Medical Center, Kansas City, Missouri, United States